CLINICAL TRIAL: NCT03076086
Title: Investigation of Secreted Phosphoproteins and PiP3 (Phosphoinositolphospat 3) in Sputum Samples of Healthy Smokers and Non Smokers
Brief Title: Investigation of Secreted Phosphoproteins and PiP3 (Phosphoinositolphospat 3) in Sputum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16-11 SPUFO I
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2017-05

CONDITIONS: Healthy; Smoking, Cigarette
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- induced sputum procedure (Experimental): Biomarker assessment (concentration of PiP3 and phosphoproteins in sputum samples) baseline and reproducibility twice in a 3 week interval of the different donors.
  Interventions: Other: Induced sputum procedure

INTERVENTIONS:
Other: Induced sputum procedure — induced sputum is a sputum specimen produced for diagnostic tests by aerosol administration of a hypertonic saline solution.

SUMMARY:
The aim of this study is to validate two new biomarkers in sputum samples. These are PiP3 (phosphoinositolphospat ) and phosphor proteins, representing important proteins within inflammatory situations of the lung.

DETAILED DESCRIPTION:
Within the study, sputum samples will be collected at 3 repetitive occasions in a 3 week interval of the different donors.

The objective is to assess for biomarker specificity and reproducibility in the two groups (smokers and non-smokers). The methods for measurement shall be validated by repetitive measurement of the sputum samples, i.e. comparison of multiple measurements of the same sample and comparison of different samples from the same donor.

ELIGIBILITY:
Inclusion Criteria:

* • Healthy male and female subjects, aged 25-45 years. Women will be considered for inclusion if they are not pregnant, as confirmed by pregnancy test and not nursing.

Females of childbearing potential need to use a highly effective method of contraception during the entire study (vasectomised partner, sexual abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the first visit until at least 72 hours after the last visit -, implants, injectables, combined oral contraceptives, hormonal IUDs (intrauterine device) or double-barrier methods, i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap).

* Body weight ≥ 50 kg and BMI (body mass index) within the range 19-32 kg/m²
* Smokers need to consume at least ten cigarettes per day and need to have at least ten packyear
* Non-smokers need to be non-smoking since at least a year with a smoking history of no more than 1 packyear.
* FEV1 (forced expiratory volume at one second)≥80% predicted and FEV1/FVC (forced expiratory vital capacity) ≥70%

Exclusion Criteria:

* • History of an acute infection four weeks prior to the informed consent visit.

  * Regular intake of medication.
  * Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis).
  * Participation in another clinical trial 30 days prior to enrollment.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Biomarker assessment | up to 3 weeks
  concentration of PiP3 and phosphoproteins in sputum samples

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hohlfeld, MD, Principal Investigator — Fraunhofer-Institute of Toxicology and Experimental Medicine
Locations (1):
- Fraunhofer ITEM, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No